CLINICAL TRIAL: NCT01999426
Title: Safety and Efficacy of Emergency On-call Respiratory Physiotherapy Services in the Paediatric Intensive Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Collaborators: Physiotherapy Research Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 05AR17; PRF/05/1 (Other Grant/Funding Number: Physiotherapy Research Foundation)
Record Dates: First submitted 2013-11-14; First posted 2013-12-03 (Estimated); Last update posted 2013-12-03 (Estimated); Status verified 2013-11

CONDITIONS: Pediatrics; Critical Care; Respiration, Artificial
Keywords: Physical Therapy Modalities; Pediatrics; Critical Care; Respiration, Artificial
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Airway clearance intervention (Experimental): Non-respiratory on-call physiotherapy treatment using airway clearance techniques
  Interventions: Other: Airway clearance intervention
- Airway clearance intervention 2 (Active Comparator): Specialist respiratory physiotherapy intervention using airway clearance techniques
  Interventions: Other: Airway clearance intervention

INTERVENTIONS:
Other: Airway clearance intervention — Both respiratory and non-respiratory on-call physiotherapists provide similar airway clearance treatments, the precise components and delivery of which will vary between physiotherapists

SUMMARY:
Emergency on-call respiratory physiotherapy cover for children in intensive care is frequently provided by physiotherapists who ordinarily work in non-respiratory areas. This has produced concerns about the safety and efficacy of on-call treatments and is widely recognised as an important clinical governance issue affecting services throughout the National Health Service (NHS).

The aim of this study is to investigate whether emergency on-call respiratory physiotherapy services provided in the paediatric intensive care unit (ICU) are safe and effective. Further it will explore whether there are any quantifiable differences between specialist and on-call physiotherapy treatments.

The study is a randomised, cross-over study design. Infants and children who are likely to require at least 2 physiotherapy treatments in one day are recruited to the study. Both physiotherapy airway clearance treatments are administered during a 12 hour period, with at least 2 hours between treatments. One is administered by a respiratory physiotherapist who works regularly in the ICU and one by a physiotherapist on the on-call rota, who normally practises in a non-respiratory clinical area. Treatments are performed in a randomised order and outcomes measured before, during and after treatments.

Physiotherapy staff who consent to participate in the study include:

Specialist respiratory physiotherapists who regularly work in the ICU Non-respiratory physiotherapists on the on-call rota who normally work in a non-respiratory areas but cover the ICU overnight and at weekends.

Patients include:

the study aims to recruit 80 infants and children (ages 0 to 16 years), who are in the paediatric intensive care unit and

1. Require full mechanical ventilation and are well sedated
2. Are likely to require at least two physiotherapy treatments within the day of the study (assessed by an independent senior respiratory physiotherapist) and
3. Whose parents or carers consent for them to participate in the study. Respiratory mechanics, arterial blood gases, oxygen saturation and peak pressures are recorded before and after each intervention Forces applied during manual techniques, flow, pressure and volume during manual lung inflations, volume of saline and selection and order of treatment components are recorded during treatments Adverse events occurring during or up to 30 minutes after physiotherapy are also recorded.

ELIGIBILITY:
Inclusion Criteria:

* infants and children who are well sedated and mechanically ventilated and likely to require at least 2 physiotherapy interventions over the course of a single day

Exclusion Criteria:

* patients in whom the application of manual techniques is contra-indicated

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 93 (Actual)
Dates: Start 2006-07; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Change in respiratory mechanics (compliance measured mL/kg/cmH2O), resistance measured in cmH2O/L/s) | 15 minutes pre- and up to 1 hour post intervention. Interventions lasted between 2 and 28 minutes)
  Respiratory compliance and resistance

SECONDARY OUTCOMES:
Force applied during manual techniques (measured in Newtons) | measured during intervention (which lasted between 2 and 28 minutes, average 8 minutes)
  Force measured during the delivery of manual techniques

OTHER OUTCOMES:
Respiratory response during intervention | measured during intervention (which lasted between 2 and 28 minutes, average 8 minutes)
  Flow (L/min), Pressure (cmH2O) and Volume (mL/kg) measured during manual lung inflations and manual techniques

CONTACTS AND LOCATIONS:
Overall Officials: Eleanor Main, PhD, Principal Investigator — University College London Institute of Child Health; Janet Stocks, PhD, Study Chair — University College London, Institute of Child Health
Locations (1):
- Great Ormond Street Hospital for Children NHS Foundation Trust, London, United Kingdom

REFERENCES:
- [Background] Shannon H, Stiger R, Gregson RK, Stocks J, Main E. Effect of chest wall vibration timing on peak expiratory fl ow and inspiratory pressure in a mechanically ventilated lung model. Physiotherapy. 2010 Dec;96(4):344-9. doi: 10.1016/j.physio.2010.02.007. Epub 2010 Apr 21. PMID 21056170
- [Background] Shannon H, Gregson R, Stocks J, Cole TJ, Main E. Repeatability of physiotherapy chest wall vibrations applied to spontaneously breathing adults. Physiotherapy. 2009 Mar;95(1):36-42. doi: 10.1016/j.physio.2008.08.004. Epub 2008 Oct 1. PMID 19627684
- [Derived] Shannon H, Stocks J, Gregson RK, Dunne C, Peters MJ, Main E. Clinical effects of specialist and on-call respiratory physiotherapy treatments in mechanically ventilated children: A randomised crossover trial. Physiotherapy. 2015 Dec;101(4):349-56. doi: 10.1016/j.physio.2014.12.004. Epub 2015 Jan 18. PMID 25749495
- [Derived] Shannon H, Stocks J, Gregson RK, Hines S, Peters MJ, Main E. Differences in delivery of respiratory treatments by on-call physiotherapists in mechanically ventilated children: a randomised crossover trial. Physiotherapy. 2015 Dec;101(4):357-63. doi: 10.1016/j.physio.2014.12.001. Epub 2015 Jan 17. PMID 25749494